CLINICAL TRIAL: NCT02330276
Title: (+)-Epicatechin: Early Phase Pre-Clinical and Initial Clinical Research on Epicatechin
Brief Title: Early Phase Pre-Clinical and Initial Clinical Research on Epicatechin
Acronym: Epicatechin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); San Diego Veterans Healthcare System (U.S. Federal Agency); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Robert R. Henry, MD, Chief, Section of Diabetes, Endocrinology and Metabolism, Veterans Medical Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08847; 1R01AT008310-01 (NIH)
Record Dates: First submitted 2014-12-23; First posted 2015-01-01 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Catechin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 10 mg (+)-epicatechin (Experimental): 4 subjects randomized to one dose of 10 mg (+)-epicatechin taken orally
  Interventions: Drug: (+)-Epicatechin
- 30 mg (+)-epicatechin (Experimental): 4 subjects randomized to one dose of 30 mg (+)-epicatechin taken orally
  Interventions: Drug: (+)-Epicatechin
- 100 mg (+)-epicatechin (Experimental): 4 subjects randomized to one dose of 100 mg (+)-epicatechin taken orally
  Interventions: Drug: (+)-Epicatechin

INTERVENTIONS:
Drug: (+)-Epicatechin — The drug to be tested is (+)-epicatechin, synthesized under GMP standards. Subjects will be given a single oral dose of (+)- epicatechin and followed on an inpatient basis over 24 hours. Three (3) different dose levels will be tested in a randomized, double-blind design: (+)- epicatechin 10 mg, 30 mg, or 100 mg. As this is a pilot study, a placebo arm will not be included.
  Other Names: Epicatechin

SUMMARY:
Early Phase Pre-Clinical and Initial Clinical Research on (+)- Epicatechin.

DETAILED DESCRIPTION:
This project is a double-blinded randomized Phase I study that will include dose-ranging one day PK and pharmacodynamic (PD) studies. Subjects will include healthy individuals and subjects who meet the American Diabetes Association (ADA) criteria for pre-diabetes, including IFG.

ELIGIBILITY:
Inclusion Criteria:

* Healthy or pre-diabetic based on medical history
* Male or female
* Must be 21 to 75 years of age (inclusive)
* Able to give informed consent to the procedures
* If female, must be either postmenopausal or test negative for pregnancy at screening and on the day of the procedure. Women on estrogen therapy will be included.
* If of childbearing potential, must practice and be willing to continue to practice appropriate birth control during the entire duration of the study
* Medication use stable for 4 weeks
* Body Mass Index (BMI) > 27 kg/m^2
* Definition of pre-diabetes: impaired fasting glucose (IFG, fasting glucose = 100-125 mg/dL) and elevated HbA1c (5.7-6.4%), each in the absence of other risk factors for diabetes

Exclusion Criteria:

* Type 2 diabetes
* Pregnancy
* Younger than 21 or older than 75 years of age
* Clinically significant abnormalities in liver or kidney function (>3x ULN), determined in the last 6 months by a certified clinical laboratory
* Recent MI or stroke (within 6 months of screening)
* Blood pressure (BP) >160 mmHg Systolic and >100 mmHg Diastolic
* Medications - thiazolidinediones, any steroids, anti-depressants, weight loss drugs
* Other diseases, besides type 2 diabetes, influencing carbohydrate metabolism

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Henry, MD, Principal Investigator — San Diego Veterans Healthcare System
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yao Q, Wei T, Qiu H, Cai Y, Yuan L, Liu X, Li X. Epigenetic Effects of Natural Products in Inflammatory Diseases: Recent Findings. Phytother Res. 2025 Jan;39(1):90-137. doi: 10.1002/ptr.8364. Epub 2024 Nov 8. PMID 39513382

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 10 mg (+)-Epicatechin | 30 mg (+)-Epicatechin | 100 mg (+)-Epicatechin
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg (+)-Epicatechin | 30 mg (+)-Epicatechin | 100 mg (+)-Epicatechin | Total
Number analyzed (Participants) | 4 | 4 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 0 | 7
  >=65 years | 1 | 0 | 4 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4
  Male | 3 | 2 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 3
  White | 0 | 4 | 4 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Circulating Urinary Concentrations of Intact Epicatechin and Epi Metabolites
Description: This will be initial PK study on synthetic (+)-epicatechin in humans. Circulating and urinary concentrations of intact epicatechin and epicatechin metabolites, including specific enantiomers
Time Frame: Baseline and 24 hours
Population: Intent to treat population (all participants who receive the medication). Last observation carried forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: nM*hr
Arm/Group | 10 mg (+)-Epicatechin | 30 mg (+)-Epicatechin | 100 mg (+)-Epicatechin
Number analyzed (Participants) | 4 | 4 | 4
nM*hr
  Metabolites (AUC nM*hr) | 105.8 (122.2) | 132.7 (148.0) | 162.3 (209.8)
  epicatechin-sulfate (AUC nM*hr) | 291.3 (119.2) | 1639 (389.0) | 3031 (1543)
  epicatechin-glucuronide (AUC nM*hr) | 3.375 (2.488) | 47.18 (39.41) | 398.3 (292.7)
  Methyl-epi-sulfate (AUC nM*hr) | 457.8 (211.5) | 3190 (496.6) | 16699 (7218)
  Total parent compound and metabolites (AUC nM*hr) | 840.3 (311.1) | 4996 (570.0) | 22563 (10335)
Statistical Analysis 1: Comparison: 10 mg (+)-Epicatechin vs 30 mg (+)-Epicatechin vs 100 mg (+)-Epicatechin; Test type: Superiority or Other; p = 0.05, General linear mixed-effects models — The reported P-Value was calculated

2. Secondary Outcome: Change From Baseline in Major Safety Endpoints
Description: Clinically significant differences in the major safety endpoints are defined as: BP (10 mm Hg change), HR (10 bpm), creatinine (>1.5 ULN), and highly conservative changes in alkaline phosphatase and liver transaminases (>1.5 ULN).
Time Frame: Baseline and 24 hours
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 10 mg (+)-Epicatechin | 30 mg (+)-Epicatechin | 100 mg (+)-Epicatechin
Number analyzed (Participants) | 4 | 4 | 4
participants | 0 | 0 | 0
Statistical Analysis 1: Comparison: 10 mg (+)-Epicatechin vs 30 mg (+)-Epicatechin vs 100 mg (+)-Epicatechin; Primary hypothesis: None of the doses of (+)-epicatechin will differ with regard to change from baseline in any of the major safety endpoints; heart rate, systolic and diastolic blood pressure; Test type: Other — one way ANOVA between groups; p < 0.05, ANOVA — for change in heart rate at 24 hr post-dosing from baseline between the 3 doses; Mean Difference (Final Values) = 77.9, 95% CI 2-sided [70.3 to 85.5], Standard Deviation 11.9

3. Secondary Outcome: Change From Baseline in Circulating Glucose Concentrations (mg/dL*24hr)
Time Frame: Baseline and 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL*24hr
Arm/Group | 10 mg (+)-Epicatechin | 30 mg (+)-Epicatechin | 100 mg (+)-Epicatechin
Number analyzed (Participants) | 4 | 4 | 4
mg/dL*24hr | 368.3 (158.5) | 342.6 (193.5) | 513.4 (185.6)
Statistical Analysis 1: Comparison: 10 mg (+)-Epicatechin vs 30 mg (+)-Epicatechin vs 100 mg (+)-Epicatechin; Test type: Superiority or Other; p = 0.05, General linear mixed-effects models — The reported P-Value was calculated

4. Secondary Outcome: Change From Baseline in Circulating Insulin Concentrations (uU/mL*24hr)
Time Frame: Baseline and 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: uU/mL*24 hr
Arm/Group | 10 mg (+)-Epicatechin | 30 mg (+)-Epicatechin | 100 mg (+)-Epicatechin
Number analyzed (Participants) | 4 | 4 | 4
uU/mL*24 hr | 1192 (488.5) | 707.2 (211.5) | 1334 (666.5)
Statistical Analysis 1: Comparison: 10 mg (+)-Epicatechin vs 30 mg (+)-Epicatechin vs 100 mg (+)-Epicatechin; Test type: Superiority or Other; p = 0.05, General linear mixed-effects models — The reported P-Value was calculated

5. Secondary Outcome: Change From Baseline in Circulating C-Peptide Concentrations (ng/mL*24hr)
Time Frame: Baseline and 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL*24hr
Arm/Group | 10 mg (+)-Epicatechin | 30 mg (+)-Epicatechin | 100 mg (+)-Epicatechin
Number analyzed (Participants) | 4 | 4 | 4
ng/mL*24hr | 61.74 (27.64) | 57.56 (28.56) | 64.23 (27.11)
Statistical Analysis 1: Comparison: 10 mg (+)-Epicatechin vs 30 mg (+)-Epicatechin vs 100 mg (+)-Epicatechin; Test type: Superiority or Other; p = 0.05, General linear mixed-effects models — The reported P-Value was calculated

ADVERSE EVENTS:
Time Frame: 9 days
Arm/Group | 10 mg (+)-Epicatechin | 30 mg (+)-Epicatechin | 100 mg (+)-Epicatechin
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg (+)-Epicatechin (N=4) | 30 mg (+)-Epicatechin (N=4) | 100 mg (+)-Epicatechin (N=4)
Intermittent Headaches (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Study subject reported having intermittent headaches (most likely due to lack of caffeine). Subject reported that the headaches resolved after taking the ibuprofen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No